CLINICAL TRIAL: NCT04694235
Title: Effect on Pregnancy Outcomes, Infant Growth and Development of an Egg Intervention During Pregnancy in Indonesia
Brief Title: Egg Intervention During Pregnancy in Indonesia
Acronym: PRECODE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Aberdeen (Other); University of Brighton (Other); University College, London (Other); Royal Veterinary College (Unknown); Birkbeck, University of London (Other); The International Livestock Research Institute (ILRI) (Other); Cheikh Anta Diop University, Senegal (Other); National Institute of Nutrition, India (Unknown); International Centre for Research in Agroforestry (Unknown); Science Made Simple (Unknown); Liverpool School of Tropical Medicine (Other); International Initiative for Impact Evaluation (Other); Digital Green Foundation (Unknown); SOAS, University of London (Unknown); University of Sheffield (Other)
Responsible Party: Principal Investigator, Dr.Umi Fahmida, Senior Researcher, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AASH Egg intervention
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Weight Gain; Anemia, Iron Deficiency; Birth Weight; Birth Length; Child Development; Zinc Deficiency; Folate Deficiency; B12 Deficiency Vitamin; Amino Acid Deficiency; Mineral Deficiency; Vitamin A Deficiency; Fatty Acid Deficiency; Parasite Infestation; E. Coli Infection; Salmonella Infections; Shigella Infection; Protozoan Infections
Keywords: Egg; Pregnancy; Indonesia; Epigenetic; Growth; Child development
MeSH Terms: conditions — Weight Gain; Anemia, Iron-Deficiency; Birth Weight; Folic Acid Deficiency; Vitamin B 12 Deficiency; Vitamin A Deficiency; Parasitic Diseases; Escherichia coli Infections; Salmonella Infections; Dysentery, Bacillary; Protozoan Infections

STUDY DESIGN:
Intervention Model Description: A total of 653 pregnant women will be recruited from 40 villages in three sub-districts. Pregnant women will be randomly allocated into the intervention or control groups. Pregnant women in the intervention group will receive boiled eggs three times per week from 2nd trimester (16-20 weeks) until delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observational cohort (control group) (No Intervention): In the observational cohort, pregnant mothers in the 2nd trimester (n=500) will be recruited and they will be followed up until their children are 24 months old. The control group women will receive standard intervention in the form of Ante Natal Care from village midwives (Polindes) or Puskesmas (IFA tablet, calcium tablet, nutrition counselling).
- Intervention group (Experimental): The intervention group women (n=153) will be provided one egg three times per week from recruitment (2nd trimester) until term along with the standard Ante Natal Care.
  Interventions: Dietary Supplement: Egg intervention

INTERVENTIONS:
Dietary Supplement: Egg intervention — Eggs are boiled until the white and yolk are firm (ca. 8 minutes) to maintain quality and safety and ensure the eggs are safe for consumption.
  Arms: Intervention group

SUMMARY:
The study consists of two arms: 1) intervention group using eggs as supplementary food given from 2nd trimester of pregnancy to birth, and 2) observational group of pregnant mothers. it aims to assess the effectiveness of improving dietary quality during pregnancy on the epigenetic and stunting related outcomes (growth and development) in infants, who will be followed up until 24 months old

DETAILED DESCRIPTION:
The study aims to assess the impact of improving dietary quality during pregnancy on the epigenetic and stunting related outcomes in infants. The open-label intervention study would be conducted alongside the observational study in the same study setting by recruitment of additional number (n=153) of pregnant women. Thus, a total of 653 pregnant women would be enrolled in the study; 153 women would be randomized to intervention arm and 500 to the control arm who would form an observational cohort of women and newborns as described above. The intervention group women will be provided one egg three times per week from recruitment (2nd trimester) until term. The control group women will receive standard intervention in the form of Ante Natal Care from village midwives or Public Health Centre (IFA tablet, calcium tablet, nutrition counselling).

ELIGIBILITY:
Inclusion Criteria:

* Woman is between 16 and 20 weeks of pregnancy based on the date of the first day of her last menstrual period.
* She is 18-40 years of age.
* She is planning to remain in the study area over the next 30 months.
* She is of Sasak ethnicity

Exclusion Criteria:

* She is expecting multiple births.
* She has a known egg allergy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 702 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stunting | birth until 24 months after delivery
  Z-score of LAZ <-2 SD based on WHO 2006
Proportion of children 10-14 months with impaired fine and gross motor skills | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess fine and gross motor skills among children aged 10 to 14 months
Proportion of children 10-14 months with impaired expressive and receptive language | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess expressive and receptive language among children aged 10 to 14 months
Proportion of children 10-14 months with impaired behavior | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess behavior among children aged 10 to 14 months
Proportion of children 10-14 months with impaired executive function | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess executive function among children aged 10 to 14 months
Proportion of children 10-14 months with impaired empathy | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess empathy among children aged 10 to 14 months
Proportion of children 10-14 months with impaired problem solving | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess problem solving among children aged 10 to 14 months
Proportion of children 10-14 months with impaired attention | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess attention among children aged 10 to 14 months
Proportion of children 10-14 months with impaired social-emotional reactivity | 10-14 months of age
  Oxford Neurodevelopment Assessment (OX-NDA) is used to assess social-emotional reactivity among children aged 10 to 14 months
Proportion of children 20-24 months with impaired motor development | 20-24 months of age
  INTERGROWTH Neurodevelopment Assessment (INTER-NDA) is used to assess motor development among children aged 20 to 24 months
Proportion of children 20-24 months with impaired cognition | 20-24 months of age
  INTERGROWTH Neurodevelopment Assessment (INTER-NDA) is used to assess cognition among children aged 20 to 24 months
Proportion of children 20-24 months with impaired language | 20-24 months of age
  INTERGROWTH Neurodevelopment Assessment (INTER-NDA) is used to assess language among children aged 20 to 24 months
Proportion of children 20-24 months with impaired social-emotional development | 20-24 months of age
  INTERGROWTH Neurodevelopment Assessment (INTER-NDA) is used to assess social-emotional development among children aged 20 to 24 months
Scores of CDI vocabulary comprehension scale in children 10-12 months | 10-12 months of age
  MacArthur-Bates Communicative Development Inventories (CDI) is used to assess vocabulary comprehension scale among children aged 10 to 12 months
Scores of CDI vocabulary production scale in children 10-12 months | 10-12 months of age
  MacArthur-Bates Communicative Development Inventories (CDI) is used to assess vocabulary production among children aged 10 to 12 months
Epigenetic state of genes associated with stunting | parents: 72 h after delivery; baby: 72 h after delivery, 24 month
  Genome-wide analysis of epigenetic states using the Illumina Infinium Methylation EPIC 850k Bead Chip (EPIC array) will be performed for selected samples from the core cohort. The outcomes will be the epigenetic state of a large number of genes which are associated with child stunting.
Epigenetic markers of birth anthropometry, adult stature, metabolic state, and cognitive ability | parents: 72 h after delivery; baby: 72 h after delivery, 24 month
  All samples (newborn, children 24 mo, parents) will be analyzed using Next Generation Bisulphite Amplicon Sequencing (BSAS) from Illumina MiSeq platform in targeted regions of the genome. The outcomes will be profiles of specific epigenetic markers of birth anthropometry, adult stature, metabolic state, and cognitive ability.

SECONDARY OUTCOMES:
Weight gain during pregnancy | 2nd trimester (16-20 weeks gestation) and 3rd trimester (28-32 weeks gestation) of pregnancy
  All measurements will be taken to the nearest 0.1 kg using standard procedures with SECA weighing machine.
Birth weight | 24 hours after birth
  All measurements will be taken to the nearest 0.1 kg using standard procedures with SECA weighing machine.
Birth length | 24 hours after birth
  All measurements will be taken to the nearest milimeter using standard procedures with SECA stadiometer/infantometer.
Hemoglobin concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their hemoglobin.
Serum ferritin concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum ferritin
Serum transferrin receptor concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum transferrin receptor
Serum zinc concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum zinc
Serum retinol concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum retinol
RBC folate concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their RBC folate
Serum vitamin B12 concentration | Mothers: second and third trimester of pregnancy
  Nutritional status measured by biochemical assessment to the mothers for their serum vitamin B12
RBC fatty acids concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their RBC fatty acids
Serum essential amino acids concentration | Mothers: second and third trimester of pregnancy
  Nutritional status measured by biochemical assessment to the mothers for their serum essential amino acids
Serum methylmalonic acid concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum methylmalonic acid
Serum choline concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum choline
Serum betaine concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum betaine
Serum vitamin B2 concentration | Mothers: second and third trimester of pregnancy
  Nutritional status measured by biochemical assessment to the mothers for their serum vitamin B2
Serum vitamin B6 concentration | Mothers: second and third trimester of pregnancy
  Nutritional status measured by biochemical assessment to the mothers for their serum vitamin B6
Serum vitamin D concentration | Mothers: second and third trimester of pregnancy
  Nutritional status measured by biochemical assessment to the mothers for their serum vitamin D
Serum CRP concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Subclinical inflammation will be measured by serum CRP in pregnant mothers and children
Serum AGP concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Subclinical inflammation will be measured by serum AGP in pregnant mothers and children
Serum RBP concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum RBP
Serum hepcidine concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum hepcidine
Serum homocysteine concentration | Mothers: second and third trimester of pregnancy; children: 6 months (+/- 2 weeks) after delivery; breastmilk: 3 and 6 months (+/- 2 weeks) after delivery
  Nutritional status measured by biochemical assessment to the mothers and children. Both the pregnant mothers and children will be measured for their serum homocysteine
Serum HbA1C concentration | Mothers: second and third trimester of pregnancy
  Gestational diabetes status will be assesed to the mothers for their serum HbA1C
Fecal myeloperoxidase (MPO) | baby: 1, 6, 24 months of age
  Gut inflammation from fecal will be measured by faecal myeloperoxidase (MPO) using ELISA
Fecal α1-antitrypsin (AAT) | baby: 1, 6, 24 months of age
  Gut inflammation from fecal will be measured by fecal α1-antitrypsin (AAT) using ELISA
Soil-transmitted helminths infection | mothers: 3rd trimester (28-32 gestational weeks) of pregnancy; baby: 1, 6, 24 months of age
  Fecal parasites from fecal will be assesed by Kato Katz and confirmed by qPCR
Bacteria infection | baby: 1, 6, 24 months of age
  Type of bacteria (Salmonella, Shigella) from fecal will be assesed by culture method
Gut microbiota | baby: 1, 6, 24 months of age
  Gut microbiota species (EPEC, ETEC, EHEC, EIEC) from fecal will be assesed using qPCR
Gut microbiome | baby: 1, 6, 24 months of age
  Faecal microbiome would be analyzed using 16S RNA sequencing of the V4 region on the Illumina MiSeq and BSAS.
Intestinal fatty acid binding protein | baby: 6 months of age
  Intestinal fatty acid binding protein from serum will be measured using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, Dr., Principal Investigator — SEAMEO RECFON
Locations (1):
- Aikmel, Sakra, and Sikur Subdistrict, Mataram, West Nusa Tenggara, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boeke CE, Gillman MW, Hughes MD, Rifas-Shiman SL, Villamor E, Oken E. Choline intake during pregnancy and child cognition at age 7 years. Am J Epidemiol. 2013 Jun 15;177(12):1338-47. doi: 10.1093/aje/kws395. Epub 2013 Feb 20. PMID 23425631
- [Background] Caudill MA, Strupp BJ, Muscalu L, Nevins JEH, Canfield RL. Maternal choline supplementation during the third trimester of pregnancy improves infant information processing speed: a randomized, double-blind, controlled feeding study. FASEB J. 2018 Apr;32(4):2172-2180. doi: 10.1096/fj.201700692RR. Epub 2018 Jan 5. PMID 29217669
- [Background] Clare CE, Brassington AH, Kwong WY, Sinclair KD. One-Carbon Metabolism: Linking Nutritional Biochemistry to Epigenetic Programming of Long-Term Development. Annu Rev Anim Biosci. 2019 Feb 15;7:263-287. doi: 10.1146/annurev-animal-020518-115206. Epub 2018 Nov 9. PMID 30412672
- [Background] Haggarty P. Epigenetic consequences of a changing human diet. Proc Nutr Soc. 2013 Nov;72(4):363-71. doi: 10.1017/S0029665113003376. Epub 2013 Sep 13. PMID 24028891
- [Background] Haggarty P, Hoad G, Campbell DM, Horgan GW, Piyathilake C, McNeill G. Folate in pregnancy and imprinted gene and repeat element methylation in the offspring. Am J Clin Nutr. 2013 Jan;97(1):94-9. doi: 10.3945/ajcn.112.042572. Epub 2012 Nov 14. PMID 23151531
- [Background] Whitelaw N, Bhattacharya S, Hoad G, Horgan GW, Hamilton M, Haggarty P. Epigenetic status in the offspring of spontaneous and assisted conception. Hum Reprod. 2014 Jul;29(7):1452-8. doi: 10.1093/humrep/deu094. Epub 2014 May 8. PMID 24812310
- [Background] Lorgen-Ritchie M, Murray AD, Ferguson-Smith AC, Richards M, Horgan GW, Phillips LH, Hoad G, Gall I, Harrison K, McNeill G, Ito M, Haggarty P. Imprinting methylation in SNRPN and MEST1 in adult blood predicts cognitive ability. PLoS One. 2019 Feb 1;14(2):e0211799. doi: 10.1371/journal.pone.0211799. eCollection 2019. PMID 30707743
- [Background] Masser DR, Stanford DR, Freeman WM. Targeted DNA methylation analysis by next-generation sequencing. J Vis Exp. 2015 Feb 24;(96):52488. doi: 10.3791/52488. PMID 25741966
- [Background] Dighe MK, Frederick IO, Andersen HF, Gravett MG, Abbott SE, Carter AA, Algren H, Rocco DA, Waller SA, Sorensen TK, Enquobahrie D, Blakey I, Knight HE, Cheikh Ismail L; International Fetal and Newborn Growth Consortium for the 21st Century. Implementation of the INTERGROWTH-21st Project in the United States. BJOG. 2013 Sep;120(Suppl 2):123-8, v. doi: 10.1111/1471-0528.12126. Epub 2013 Jul 11. PMID 23841827
- [Background] Weisenberger D, Van Den Berg D, Pan F, Berman B, Laird P. Comprehensive DNA methylation analysis on the Illumina Infinium assay platform. Illumina, San Diego. 2008.
- [Background] Fenson L, Pethick S, Renda C, Cox JL, Dale PS, Reznick JS. Short-form versions of the MacArthur communicative development inventories. Applied Psycholinguistics. 2000;21(1):95-116.
- [Background] Zeisel SH, Mar MH, Howe JC, Holden JM. Concentrations of choline-containing compounds and betaine in common foods. J Nutr. 2003 May;133(5):1302-7. doi: 10.1093/jn/133.5.1302. PMID 12730414
- [Background] Patterson KY, Bhagwat SA, Williams JR, Howe JC, Holden J, Zeisel S, et al. USDA database for the choline content of common foods, release two. Nutrient Data Laboratory, Beltsville Human Nutrition Research Center, ARS, USDA. 2008.
- [Background] Cho E, Zeisel SH, Jacques P, Selhub J, Dougherty L, Colditz GA, Willett WC. Dietary choline and betaine assessed by food-frequency questionnaire in relation to plasma total homocysteine concentration in the Framingham Offspring Study. Am J Clin Nutr. 2006 Apr;83(4):905-11. doi: 10.1093/ajcn/83.4.905. PMID 16600945
- [Background] Mhila G, DeRenzi B, Mushi C, Wakabi T, Steele M, Dhaldialla P, et al. Using mobile applications for community-based social support for chronic patients. Health Informatics in Africa. 2009.
- [Background] Sethi V, Tiwari K, Sareen N, Singh S, Mishra C, Jagadeeshwar M, Sunitha K, Kumar SV, de Wagt A, Sachdev HPS. Delivering an Integrated Package of Maternal Nutrition Services in Andhra Pradesh and Telangana (India). Food Nutr Bull. 2019 Sep;40(3):393-408. doi: 10.1177/0379572119844142. Epub 2019 Jun 16. PMID 31204503
- [Background] Lutter CK, Iannotti LL, Stewart CP. Cracking the egg potential during pregnancy and lactation. Sight Life. 2016;30:75-81.
- [Background] Jacobson SW, Carter RC, Molteno CD, Stanton ME, Herbert JS, Lindinger NM, Lewis CE, Dodge NC, Hoyme HE, Zeisel SH, Meintjes EM, Duggan CP, Jacobson JL. Efficacy of Maternal Choline Supplementation During Pregnancy in Mitigating Adverse Effects of Prenatal Alcohol Exposure on Growth and Cognitive Function: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Alcohol Clin Exp Res. 2018 Jul;42(7):1327-1341. doi: 10.1111/acer.13769. Epub 2018 Jun 15. PMID 29750367
- [Background] Yan J, Jiang X, West AA, Perry CA, Malysheva OV, Devapatla S, Pressman E, Vermeylen F, Stabler SP, Allen RH, Caudill MA. Maternal choline intake modulates maternal and fetal biomarkers of choline metabolism in humans. Am J Clin Nutr. 2012 May;95(5):1060-71. doi: 10.3945/ajcn.111.022772. Epub 2012 Mar 14. PMID 22418088